CLINICAL TRIAL: NCT00494195
Title: Phase I Gene Transfer of rAAV1.tMCK.Human-alpha-sarcoglycan for Limb Girdle Muscular Dystrophy Type 2D (LGMD2D)
Brief Title: Gene Transfer Therapy for Treating Children and Adults With Limb Girdle Muscular Dystrophy Type 2D (LGMD2D)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Muscular Dystrophy Association (Other)
Responsible Party: Principal Investigator, Jerry R. Mendell, Director, Center for Gene Therapy, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5U54AR050733 (NIH); U54AR050733 (NIH); 5U54AR050733 (NIH); IRB07-00329
Record Dates: First submitted 2007-06-27; First posted 2007-06-29 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Muscular Dystrophies
Keywords: limb girdle muscular dystrophy type 2D; alpha-sarcoglycanopathy; LGMD; LGMD2D; gene therapy; gene transfer; muscular dystrophy; SGCA; sarcoglycan; limb girdle; adeno-associated virus; AAV; AAV1
MeSH Terms: conditions — Muscular Dystrophies; Sarcoglycanopathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): The first cohort will receive a total of 1.5 ml volume of study agent in two to six separate injections into the selected muscle (extensor digitorum brevis) or other muscle if more appropriate upon considering the individual patient. The dose will be 3.25 X 10 to the 11 vg in 1.5 ml. The anatomical midline point of the muscle will be identified on the skin and two to six vector injections will be distributed in the direction of an X. In each cohort, only one extremity will receive vector with transgene while the opposite extremity will be injected with placebo.
  Interventions: Genetic: rAAV1.tMCK.human-alpha-sarcoglycan- First cohort
- 2 (Experimental): The second cohort will receive the same dose of 3.25 X 10 to the 11 vg in 1.5 ml delivered to muscle according to the same paradigm. In each cohort, only one extremity will receive vector with transgene while the opposite extremity will be injected with placebo.
  Interventions: Genetic: Genetic: rAAV1.tMCK.human-alpha-sarcoglycan- Second cohort

INTERVENTIONS:
Genetic: rAAV1.tMCK.human-alpha-sarcoglycan- First cohort — The first cohort of subjects with LGMD2D (alpha-sarcoglycan deficiency) and proven mutations will undergo gene transfer with a minimum of three subjects enrolled into this cohort and will receive a total of 1.5 ml volume of study agent in two to six separate injections into the selected muscle (extensor digitorum brevis) or other muscle if more appropriate upon considering the individual patient. The dose will be 3.25 X 10 to the 11 vg in 1.5 ml.
  In each cohort, only one extremity will receive vector with transgene while the opposite extremity will be injected with placebo.
  Other Names: LGMD2D Gene therapy-First cohort
  Arms: 1
Genetic: Genetic: rAAV1.tMCK.human-alpha-sarcoglycan- Second cohort — The second cohort will receive the same dosis of 3.25 X 10 to the 11 vg in 1.5 ml delivered to muscle according to the same paradigm. In each cohort, only one extremity will receive vector with transgene while the opposite extremity will be injected with placebo.
  Other Names: LGMD2D Gene therapy- Second cohort
  Arms: 2

SUMMARY:
Limb girdle muscular dystrophy type 2D (LGMD2D) is a genetic disease that affects skeletal muscle. Insufficient levels of the protein alpha-sarcoglycan result in muscle weakness that worsens over time. The purpose of this study is to evaluate the safety and effectiveness of gene therapy in treating children and adults with LGMD2D.

DETAILED DESCRIPTION:
The primary objective of this study is the assessment of the safety of intramuscular administration to alpha-sarcoglycan deficient subjects of recombinant adeno-associated virus serotype 1 (rAAV1)-human alpha-sarcoglycan gene (hαSG) vector under control of a skeletal muscle creatine kinase promoter. The secondary objective is to determine the dose of rAAV1.tMCK.hαSG vector required to achieve a detectable level of alpha-sarcoglycan in muscle of subjects with this disorder.

A recombinant virus vector constructed from AAV1 has been altered to carry the human alpha-sarcoglycan gene expressed from a tMCK promoter. The construct has been shown to initiate the production of a functional alpha-sarcoglycan protein in laboratory animals. This construct can reverse the dystrophic phenotype in the alpha-sarcoglycan knock out mouse, a laboratory animal model for the clinical disorder. Intramuscular injection of rAAV1 restores muscle histology to normal and increases muscle strength to levels exceeding control knock out mice but not to the same degree as wild-type mice.

The proposed human clinical trial is a phase I, double-blind randomized protocol with injection of rAAV1.tMCK.hαSG gene vector into muscle. Two cohorts of subjects with LGMD2D(alpha-sarcoglycan deficiency), each with proven mutations will undergo gene transfer. A minimum of three subjects will be enrolled into each cohort. The first cohort will receive a total of 1.5 ml volume of study agent in two to six separate injections into the selected muscle (extensor digitorum brevis) or other muscle if more appropriate considering the individual patient) with a dose of 3.25 X 10 to the 11 vg in 1.5 ml. The anatomical midline point of the muscle will be identified on the skin and 2 to 6 vector injections will be distributed in the direction of an X. The second cohort will receive the same dose delivered to muscle according to the same paradigm. In each cohort, only one extremity will receive vector with transgene while the opposite extremity will be injected with placebo. On the day of the vector infusion, 4 hours before gene transfer, patients will receive intravenous methylprednisolone 2.0 mg/kg (not to exceed 1 gm total), with repeat doses on two consecutive mornings. The methylprednisolone is specifically given to diminish the immediate inflammation from the needle injection, which is known to arouse an inflammatory reaction and could contribute to bringing antigen presenting cells to the site of vector delivery. We have previously demonstrated that this treatment enhances gene expression by at least 2-fold (Included as part of BB-IND-12936 for minidystrophin gene transfer).

Safety endpoints to be assessed include inflammatory reaction to the vector, as evaluated by muscle biopsy, and changes in hematology, serum chemistry, urinalysis, immunologic responses to rAAV1 and alpha-sarcoglycan, and reported history and observations of symptoms. The patient will have 10 to 12 follow-up visits for the next 2 years after the initial infusion.

ELIGIBILITY:
Inclusion Criteria:

* Six LGMD2D subjects ages 5 and older based on the clinical degree of involvement (impaired muscle function/weakness, sufficient muscle preservation)
* Preservation of EDB muscle or another muscle if judged more favorable because of adequate muscle mass for gene transfer
* Males and females of any ethnic group
* Established mutations of an -SG gene on both alleles
* Ability to cooperate for testing
* Sexually active patients must be willing to practice a reliable method of contraception during the study

Exclusion Criteria:

* Active viral infection (symptoms listed in section 9.0 of the protocol)
* LGMD2D subjects without weakness or functional loss
* Cardiomyopathy based on clinical exam and ECHO with ejection fraction less than 40%
* HIV infected
* Hepatitis A, B, or C infected
* Autoimmune diseases and immunosuppressive drugs (other than pulse methylprednisolone at time of gene transfer)
* Persistent leucopenia or leucocytosis (WBC less than or equal to 3.5 K/cu mm or at least 20.0 K/ cu mm) or neutrophils less than 1.5 K/ cu mm
* Concomitant illness or requirement for chronic drug treatment that in the opinion of the Principal Investigator creates unnecessary risks for gene transfer
* Pregnancy
* Abnormal laboratory values considered clinically significant
* Alcoholism (CAGE questionnaire), and laboratory tests such as GGT and MCV

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-03; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Safety of AAV1.tMCK.human-alpha-sarcoglycan gene transfer via intramuscular injection to the EDB muscle | Measured throughout the study

SECONDARY OUTCOMES:
Human-alpha-sarcoglycan gene expression at the site of gene transfer via muscle biopsy | First cohort: Measured 45 days for two patients and at 90 days after gene transfer for one patient; Second cohort: Measured at 6 months after gene transfer for the three patients
Muscle strength of the gene transferred muscle via maximal volume isometric contraction testing (MVICT) if selected muscle is suitable for strenght testing | Measured 45 or 90 days after gene transfer in the first cohort, or 6 months post-gene transfer in second cohort depending on muscle biopsy date

CONTACTS AND LOCATIONS:
Overall Officials: Jerry R. Mendell, MD, Principal Investigator — The Research Institute at Nationwide Children's Hospital
Locations (1):
- The Research Institute at Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] Allamand V, Donahue KM, Straub V, Davisson RL, Davidson BL, Campbell KP. Early adenovirus-mediated gene transfer effectively prevents muscular dystrophy in alpha-sarcoglycan-deficient mice. Gene Ther. 2000 Aug;7(16):1385-91. doi: 10.1038/sj.gt.3301247. PMID 10981665
- [Background] Buning H, Nicklin SA, Perabo L, Hallek M, Baker AH. AAV-based gene transfer. Curr Opin Mol Ther. 2003 Aug;5(4):367-75. PMID 14513679
- [Background] Bueno MR, Moreira ES, Vainzof M, Chamberlain J, Marie SK, Pereira L, Akiyama J, Roberds SL, Campbell KP, Zatz M. A common missense mutation in the adhalin gene in three unrelated Brazilian families with a relatively mild form of autosomal recessive limb-girdle muscular dystrophy. Hum Mol Genet. 1995 Jul;4(7):1163-7. doi: 10.1093/hmg/4.7.1163. PMID 8528203
- [Background] Rodino-Klapac LR, Lee JS, Mulligan RC, Clark KR, Mendell JR. Lack of toxicity of alpha-sarcoglycan overexpression supports clinical gene transfer trial in LGMD2D. Neurology. 2008 Jul 22;71(4):240-7. doi: 10.1212/01.wnl.0000306309.85301.e2. Epub 2008 Jun 4. PMID 18525034
- [Result] Mendell JR, Rodino-Klapac LR, Rosales XQ, Coley BD, Galloway G, Lewis S, Malik V, Shilling C, Byrne BJ, Conlon T, Campbell KJ, Bremer WG, Taylor LE, Flanigan KM, Gastier-Foster JM, Astbury C, Kota J, Sahenk Z, Walker CM, Clark KR. Sustained alpha-sarcoglycan gene expression after gene transfer in limb-girdle muscular dystrophy, type 2D. Ann Neurol. 2010 Nov;68(5):629-38. doi: 10.1002/ana.22251. PMID 21031578
- [Result] Mendell JR, Rodino-Klapac LR, Rosales-Quintero X, Kota J, Coley BD, Galloway G, Craenen JM, Lewis S, Malik V, Shilling C, Byrne BJ, Conlon T, Campbell KJ, Bremer WG, Viollet L, Walker CM, Sahenk Z, Clark KR. Limb-girdle muscular dystrophy type 2D gene therapy restores alpha-sarcoglycan and associated proteins. Ann Neurol. 2009 Sep;66(3):290-7. doi: 10.1002/ana.21732. PMID 19798725
- See also: Click here for the Nationwide Children's Hospital Web site — http://www.nationwidechildrens.org/center-for-gene-therapy
- See also: Click here for the Muscular Dystrophy Association Web site — http://www.mdausa.org